CLINICAL TRIAL: NCT07102043
Title: Glucose Metabolism in CFRD: Exploring the Role of CFTR Modulators in Metabolic Dysfunction
Brief Title: Glucose Metabolism in Cystic Fibrosis Related Diabetes (CFRD)
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rita Basu, Endowed Professor of Diabetes Science; Medical Director, Office of Human Research Protection Program, and Chair of the Institutional Review Board, University of Alabama at Birmingham
Other Study IDs: IRB300014949; P30DK072482 (NIH)
Record Dates: First submitted 2025-06-17; First posted 2025-08-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis Related Diabetes
Keywords: Cystic Fibrosis Related Diabetes; cystic fibrosis transmembrane conductance regulator (CFTR); CFTR modulators; Elexacaftor/ tezacaftor/ivacaftor or ETI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Participant biospecimen will be retained until all analysis for outcome measures are complete and results published. DNA will not be extracted retained samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CFRD F508del +ETI: CFRD with at least one copy of F508del currently on elexacaftor/tezacaftor/ivacaftor (CFRDF508del+ETI),
- CFRD-ETI: CFRD with a mutation that is not eligible for modulator therapy (CFRD-ETI).

SUMMARY:
The study aims to test whether use of CFTR modulators (ETI) improves fasting and post prandial glycemia by enhancing disposition index (DI) in individuals with CFRD with CFTR +ve mutation (at least one copy of F508del) on CFTR modulator (ETI) therapy (CFRDF508del+ETI). CFRD with a mutation that is not eligible for modulator therapy (CFRD-ETI) will be the control group.

DETAILED DESCRIPTION:
This is a mechanistic observational study. A physiological challenge of a single mixed meal tolerance test (MMTT) is administered, which will enable a comprehensive assessment of multiple parameters of glucose turnover, insulin secretion, insulin sensitivity and lipolysis in individuals with CFRD. The MMTT is the gold standard for measuring both insulin action and secretion simultaneously with glucose kinetics. The pilot study aims to test whether use of CFTR modulators (ETI) improves fasting and post prandial glycemia by enhancing disposition index (DI) in individuals with CFRD with CFTR +ve mutation (at least one copy of F508del) on CFTR modulator (ETI) therapy (CFRDF508del+ETI).

We plan to gather critical preliminary data on the following aspects of CFRD:

1. Abnormalities in specific components (basal vs. static vs. dynamic) of beta-cell function in CFRDF508del+ETI and in CFRD-ETI individuals.
2. Effects of ETI on components of beta cell function.
3. Effects of CFTR mutation and of CFTR modulators (CFRDF508del+ETI) on insulin sensitivity and post prandial glucose turnover in CFRD.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have at least one copy of the F508 deletion and are on ETI medications and individuals who have a different mutation and are not eligible for ETI medications
* Age 21-75 years at time of consent
* BMI 19-50 kg/m2 (In Asians BMI is ~ 2 points lower for comparison so it is 17-48 kg/m2)
* Creatinine ≤ 1.4 mg/dl in women and ≤ 1.5 mg/dl in men
* HbA1c ≤ 11% lifestyle treatment or mono/combination therapy with oral hypoglycemic agents (e.g. metformin or sulphonylurea or SGLT2i) and/or insulin.
* Willing to be at a stable weight for duration of the study.
* An understanding of and willingness to follow the protocol and sign the informed consent

Exclusion Criteria:

* Debilitating chronic disease
* Anemia <10 gm/dL in females and <11.0 gm/dL in males
* Symptoms of undiagnosed illness on history/exam
* Abuse of alcohol or recreational drugs
* Pregnancy
* Active hepatic disease
* Current use of the following drugs and supplements: corticosteroids, benzodiazepines, opiates, barbiturates, anticoagulant therapy
* Any other medication that the investigator believes is a contraindication to the subject's participation

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Cystic Fibrosis related Diabetes (CFRD)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Disposition Index in CFRD | Day 1 During the Mixed meal test
  Disposition Index (DI - β-cell responsivity appropriate to the degree of insulin resistance) is higher in CFRDF508del+ETI when compared to CFRD with a mutation not eligible to be on ETI (CFRD-ETI).

SECONDARY OUTCOMES:
Post prandial glucose turnover | Day 1 During the mixed meal test
  Post prandial glucose turnover is improved in CFRDF508del+ETI when compared to CFRD with a mutation not eligible to be on ETI (CFRD-ETI).

CONTACTS AND LOCATIONS:
Overall Officials: Rita Basu, MD, Principal Investigator — UAB Medicine
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared, however cumulative data from all participants will be made available on completion of study as per NIH data sharing policy.